CLINICAL TRIAL: NCT03949478
Title: An Initial Clinical Study to Treat Postictal Symptoms
Brief Title: Treating Postictal Symptoms Using Ibuprofen and Nifedipine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPS-1.0
Record Dates: First submitted 2019-04-11; First posted 2019-05-14 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Epilepsy; Epilepsies, Partial
Keywords: Postictal; Blood flow
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial | interventions — Ibuprofen; Nifedipine

STUDY DESIGN:
Intervention Model Description: We will study 90 subjects admitted to hospital for epilepsy investigations. We will randomly divide the patients into three treatment groups (30 patients each). They will receive either placebo, ibuprofen, or nifedipine while in hospital. We will then determine the effect of each of these treatments on the severity of hypoperfusion and neurological deficits that follows their seizures.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The UofC Clinical Research Unit, which has no contact with patients or clinicians, will prepare the concealed randomization schedule and the randomization tool. Our research pharmacy will prepare three identical tablets to be given to each subject. The participant, care provider, investigators, and outcomes assessors will be blinded to treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Patients will receive placebo for at least five days prior to the first blood flow study. They will continue to receive placebo until the baseline study is obtained after the postictal study has been completed.
  Interventions: Drug: Placebo
- Ibuprofen (Experimental): Patients will receive ibuprofen 400 mg by mouth three times a day (po tid) for at least five days prior to the first blood flow study. They will continue to receive ibuprofen until the baseline study is obtained after the postictal study has been completed.
  Interventions: Drug: Ibuprofen
- Nifedipine (Experimental): Patients will receive nifedipine 10 mg po tid for 2 days, then 20 mg po tid, thereafter for at least five days prior to the first blood flow study. They will continue to receive nifedipine until the baseline study is obtained after the postictal study has been completed.
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen to be prepared in a tablet that is not distinguishable from nifedipine or placebo tablet.
  Other Names: Advil headache & migraine extra strength; DIN 02467658
  Arms: Ibuprofen
Drug: Nifedipine — Nifedipine to be prepared in a tablet that is not distinguishable from ibuprofen or placebo tablet.
  Other Names: Adalat XL 20 mg, DIN 02237618; Adalat XL 30 mg, DIN 02155907
  Arms: Nifedipine
Drug: Placebo — Sugar pill to be prepared in a tablet that is not distinguishable from ibuprofen or nifedipine tablet.
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of ibuprofen or nifedipine on post-seizure hypoperfusion and neurological deficits in patients with epilepsy. One group will receive ibuprofen, another will receive nifedipine, and anther placebo.

DETAILED DESCRIPTION:
Immediately following seizures, brain blood flow is significantly reduced for approximately one hour and is located to the brain area where the seizure originated. This may contribute to symptoms that patients experience immediately following seizures and in between seizures.

Animal studies have shown that that giving anti-inflammatory drugs (e.g., ibuprofen) and blood pressure medications (e.g., nifedipine) prevents the hypoperfusion and behavioural impairments seen in animals immediately following seizures. Thus, two classes of inexpensive and well-tolerated drugs - already in clinical use - have been identified that can be tested in humans to prevent the serious consequences that follow seizures.

The investigators will study 90 subjects admitted to hospital for epilepsy investigations. The investigators will randomly divide the patients into three treatment groups (30 patients each). Patients will receive either placebo, ibuprofen, or nifedipine while in hospital. The effect of each of these treatments on the severity of hypoperfusion and neurological deficits that follows seizures will then be assessed.

ELIGIBILITY:
Inclusion Criteria:

* age > 16 yrs, frequent seizures (>1 per week) and cognitive ability sufficient to complete neuropsychological testing.

Exclusion Criteria:

* multiple seizure onset zones, contraindications to CT or MR imaging, any contraindication to ibuprofen or nifedipine, as well as current or recent (< 2 months) exposure COX-2 inhibitor or calcium channel blocker.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Postictal blood flow | 5 - 40 days
  Change in cerebral blood flow following seizures, relative to baseline. It will be measured by CT perfusion or ASL MRI.

SECONDARY OUTCOMES:
Neuropsychological performance - Picture Sequence Memory Test | 5 - 40 days
  For all Cognition Domain tests, three standardized scores are provided:
  * An uncorrected score comparing the test-taker to all individuals in the NIH Toolbox normative sample (mean = 100, SD = 15);
  * An age-corrected score that compares the test-taker to NIH Toolbox age-matched individuals (mean = 100, standard deviation = 15); and
  * A fully-corrected T-score that adjusts for key demographic variables including age, sex, race/ethnicity, and educational attainment (mean = 50, standard deviation = 10).
  Measure = Picture sequence memory Construct = Episodic memory
  Scale ranges:
  * uncorrected score (mean = 100, SD = 15).
  * age-corrected score (mean = 100, SD = 15).
  * fully-corrected T-score (mean = 50, SD = 10). For this test, a greater standardized score indicates better episodic memory.
Neuropsychological performance - Flanker Inhibitory Control and Attention Test | 5 - 40 days
  Measure = Flanker Inhibitory Control and Attention Test Construct = Executive Function & Attention
  Scale ranges:
  * uncorrected score (mean = 100, standard deviation = 15). Higher score is better
  * age-corrected score (mean = 100, standard deviation = 15). Higher score is better.
  * fully-corrected T-score (mean = 50, standard deviation = 10). Higher score is better.
  For this test, a higher raw or standardized score indicates greater inhibitory control and attention.
Neuropsychological performance - List Sorting Working Memory Test | 5 - 40 days
  Measure = List Sorting Working Memory Test Construct = Working Memory
  Scale ranges:
  * uncorrected score (mean = 100, standard deviation = 15). Higher score is better
  * age-corrected score (mean = 100, standard deviation = 15). Higher score is better.
  * fully-corrected T-score (mean = 50, standard deviation = 10). Higher score is better.
  For this test, a greater raw or standardized score indicates better episodic memory.
Neuropsychological performance - Picture Vocabulary Test | 5 - 40 days
  Measure = Picture Vocabulary Test Construct = Language
  Scale ranges:
  * uncorrected score (mean = 100, standard deviation = 15). Higher score is better
  * age-corrected score (mean = 100, standard deviation = 15). Higher score is better.
  * fully-corrected T-score (mean = 50, standard deviation = 10). Higher score is better.
  For this test, a higher standardized score indicates greater general vocabulary knowledge.
Neuropsychological performance- Oral Reading Recognition Test | 5 - 40 days
  Measure = Oral Reading Recognition Test Construct = Language
  Scale ranges:
  * uncorrected score (mean = 100, standard deviation = 15). Higher score is better
  * age-corrected score (mean = 100, standard deviation = 15). Higher score is better.
  * fully-corrected T-score (mean = 50, standard deviation = 10). Higher score is better.
  For this test, a higher standardized score indicates a greater ability to read aloud.
Neuropsychological performance - Dimensional Change Card Sort Test | 5 - 40 days
  Measure = Dimensional Change Card Sort Test Construct = Executive function
  Scale ranges:
  * uncorrected score (mean = 100, standard deviation = 15). Higher score is better
  * age-corrected score (mean = 100, standard deviation = 15). Higher score is better.
  * fully-corrected T-score (mean = 50, standard deviation = 10). Higher score is better.
  For this test, a greater raw or standardized score indicates greater cognitive flexibility.
Neuropsychological performance - Pattern Comparison Processing Speed Test | 5 - 40 days
  Measure = Pattern Comparison Processing Speed Test Construct = Processing Speed
  Scale ranges:
  * uncorrected score (mean = 100, standard deviation = 15). Higher score is better
  * age-corrected score (mean = 100, standard deviation = 15). Higher score is better.
  * fully-corrected T-score (mean = 50, standard deviation = 10). Higher score is better.
  For this test, a greater raw or standardized score indicates faster processing speed.
Psychological well-being | 5 - 40 days
  The Psychological Well-Being measure assesses a subjective and experiential aspect of pleasure and positive affect, as well as fulfillment and purpose. Psychological Well-being composite scores are generated as the weighted average of the uncorrected standardized score (T scores; mean = 50, SD = 10) obtained from each subdomain:
  Positive Affect Construct = This portion assesses positive affect, or feelings of a pleasurable engagement with the environment, using a positive affect survey.
  Higher scores = more positive affect.
  Life Satisfaction Construct = This portion assesses how the participant evaluates their life, in terms of whether they like it or not, using a life satisfaction survey.
  Higher scores = greater life satisfaction.
  Meaning and Purpose Construct = This portion evaluates the degree to which the participant feels their life matters or makes sense.
  Higher scores = greater sense of meaning and purpose.
Social Relationships | 5 - 40 days
  The Social Relationships measure assesses the participants social network structure, extent, and quality. Composite social satisfaction composite scores are generated as the weighted average of the T-scores (mean = 50, SD = 10) from the subdomains, with loneliness and perceived rejection reverse-coded.
  Perceived Social Support Construct = This portion evaluates the degree to which the participant feels their life matters or makes sense.
  Higher scores = greater sense of meaning and purpose.
  Companionship Construct = This portion assesses self-reported perceptions of the participant has companions to interact with and perceptions of being alone or lonely.
  Higher scores = higher perceived friendship or more loneliness.
  Social Distress Construct = This portion evaluates the degree to which the participant feels their life matters or makes sense.
  Higher scores = greater perceived hostility and rejection.
Stress and Self-Efficacy Relationships | 5 - 40 days
  The Stress and Self-Efficacy measure assesses the individual's perception of life events and their relationships as well as their perceived coping skills. Stress and self-efficacy composite scores are generated as the weighted average of the T-scores (mean = 50, SD = 10) from the subdomains
  Perceived Stress Construct = This portion evaluates the participants perceived stress. Higher scores = greater perceived stress.
  Self-Efficacy Construct = This portion assesses self-efficacy, or the participants belief in their capacity to manage and have control over events.
  Higher scores = more general self-efficacy.
Negative affect | 5 - 40 days
  composite scores are generated as the weighted average of the T-scores from the subdomains. Negative affect includes the following subdomains:
  Anger Construct = This portion assesses attitudes of hostility and cynicism. Higher scores = higher levels of anger.
  Fear Construct = This portion assesses the participants perception of threat and autonomic arousal associated with fear.
  Higher scores = higher levels of fear.
  Sadness Construct = This portion assesses the participants feelings of sadness, or their low levels of positive affect or low mood.
  Higher scores = more sadness.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Federico, MD, PhD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - South Health Campus, Calgary, Alberta